CLINICAL TRIAL: NCT01388504
Title: Does Sodium Nitrite Administration Reduce Ischaemia-reperfusion Injury in Patients Presenting With Acute ST Segment Elevation Myocardial Infarction?
Brief Title: Nitrites in Acute Myocardial Infarction
Acronym: NIAMI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government); Medical Research Council (Other Government); St George's Healthcare NHS Trust (Other); Brighton and Sussex University Hospitals NHS Trust (Other); Imperial College London (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3/030/10
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-11

CONDITIONS: Acute ST Elevation Myocardial Infarction
MeSH Terms: interventions — Sodium Nitrite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sodium nitrite (Experimental)
  Interventions: Drug: sodium nitrite
- placebo (Placebo Comparator): sterile solution containing 0.9%w/v sodium chloride in 5ml water injected intravenously over a period of 2½ - 5 minutes
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: sodium nitrite — sterile solution containing low dose sodium nitrite dissolved in 5ml water injected intravenously over a period of 2½ - 5 minutes immediately prior to opening of the infarct related artery using Percutaneous Coronary Intervention
  Arms: sodium nitrite
Other: Placebo — sterile solution containing 0.9%w/v sodium chloride in 5ml water injected intravenously over a period of 2½ - 5 minutes immediately prior to Percutaneous Coronary Intervention
  Arms: placebo

SUMMARY:
The research question to be addressed is "Does a 2.5 - 5 minute systemic intravenous injection of sodium nitrite administered immediately before opening of the infarct related artery result in significant reduction of ischaemia reperfusion injury in patients with first acute ST elevation myocardial infarction (MI)?"

DETAILED DESCRIPTION:
There are estimated to be 125,000 acute myocardial infarctions (heart attacks) in the UK every year. Although substantial progress has been made in reducing the infarct size by prompt opening of the infarct related artery (with thrombolytic therapy or percutaneous coronary intervention (PCI)), effective therapy to further reduce the infarct size would substantially reduce the risk of the patient subsequently developing heart failure.

There is a growing body of evidence from studies in animals that the use of nitrites may help in reducing the infarct size, although this has not been tested in man.

In this phase 2/3 study, the investigators propose to investigate the effect of sodium nitrite injection on infarct size. Eligible patients will be males aged 18 and over and females aged 55 and over, presenting within 12 hours of the onset of chest pain, who are suitable for treatment with percutaneous coronary intervention. Those who give verbal agreement to take part will receive a 2.5-5 minute injection of sodium nitrite (or placebo) immediately prior to the blocked artery being opened with percutaneous coronary intervention.

ELIGIBILITY:
Men aged ≥18 years, women aged ≥55 years, and women <55years who are sterilised, or have had a hysterectomy or have effective contraception and thus where there is no possibility of them being pregnant; presenting within 12 hours of the onset of chest pain who have ST segment elevation of more than 1mm elevation in limb leads or 2mm elevation in two contiguous chest leads or new left bundle branch block (LBBB) and for whom the clinical decision has been made to treat with primary PCI will be eligible for enrolment. Occlusion of the culprit related artery (TIMI grade 0 or TIMI grade 1) will also be required for inclusion. Eligible patients will be of North European descent.

Exclusion criteria

* Historical or ECG evidence of previous myocardial infarction
* Patients with prior coronary artery bypass grafting (CABG)
* Prior revascularization procedure where this procedure (PCI) was performed in the same territory as the current infarct
* Known or suspected pregnancy
* Contra-indications to MRI
* Patients with cardiac arrest or cardiogenic shock
* Patients with left main coronary occlusion
* Patients with known moderate to severe renal failure (estimated GFR < 30mls/min), or liver failure
* Patients with prior thrombolysis for this event
* Patients with such Left Main disease which after PCI of their culprit lesion (culprit lesions may be located in the LAD or LCx or RCA) are likely to require CABG within the time course of the study period (6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Infarct size corrected for area at risk (using ESA) | 6-8 days post injection

SECONDARY OUTCOMES:
Left ventricular ejection fraction and end systolic volume index | 6-8 days and 6 months post injection
Plasma creatine kinase | 72 hours post injection
Troponin I | 72 hours post injection
Infarct size corrected for area at risk | 6 months
Infarct size corrected for area at risk (using T2) | 6-8 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frenneaux, MD, FRCP, Study Director — University of Aberdeen; Juan Carlos Kaski, MD, FRCP, Principal Investigator — St George's Healthcare NHS Trust; David HildickSmith, MD, FRCP, Principal Investigator — Brighton and Sussex University Hospitals NHS Trust
Locations (3):
- United Kingdom (3):
  - Aberdeen Royal Infirmary, Aberdeen
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - St George's Healthcare NHS Trust, London

REFERENCES:
- [Derived] Siddiqi N, Bruce M, Neil CJ, Jagpal B, Maclennon G, Cotton SC, Papadopoulo SA, Bunce N, Lim P, Schwarz K, Singh S, Hildick-Smith D, Horowitz JD, Madhani M, Boon N, Kaski JC, Dawson D, Frenneaux MP. Protocol: does sodium nitrite administration reduce ischaemia-reperfusion injury in patients presenting with acute ST segment elevation myocardial infarction? Nitrites in acute myocardial infarction (NIAMI). J Transl Med. 2013 May 6;11:116. doi: 10.1186/1479-5876-11-116. PMID 23648219